CLINICAL TRIAL: NCT03459443
Title: An Open-Label Phase 2 Proof-of-Concept Study in Patients With C3 Glomerulopathy (C3G) or Immune-Complex Membranoproliferative Glomerulonephritis (IC-MPGN) Treated With ACH-0144471
Brief Title: A Proof of Concept Study for a 12 Month Treatment in Patients With C3G or IC-MPGN Treated With ACH-0144471
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason for terminating study early was inconclusive efficacy results. No safety findings were identified.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH471-205; 2017-002674-39 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: C3 Glomerulonephritis; C3 Glomerulopathy; Immune Complex Membranoproliferative Glomerulonephritis; IC-MPGN; Dense Deposit Disease
Keywords: factor D; fD; alternative pathway; complement mediated disease; C3GN; DDD; idiopathic MPGN; MPGN Type I; MPGN Type II; MPGN Type III; Primary MPGN; MCGN; Mesangiocapillary Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — danicopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Danicopan (Experimental): Danicopan was to be administered to participants with C3G or IC-MPGN at a starting dose of 100 milligrams (mg) 3 times daily (TID) for the first 2 weeks, then the dosage was to be increased to 200 mg TID for the remainder of the study.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Danicopan was to be administered as an oral tablet.
  Other Names: ACH-4471; ACH4471; 4471; ALXN2040

SUMMARY:
The primary purpose of this study was to evaluate the efficacy of 12 months of oral ACH-0144471 (also known as danicopan and ALXN2040) in participants with C3G or IC-MPGN based on histologic scoring and proteinuria.

DETAILED DESCRIPTION:
This was an open-label study to evaluate the efficacy of treatment with danicopan in participants 12 years of age or older with biopsy-confirmed C3G or IC-MPGN who had not undergone renal transplantation. All participants were to receive active treatment with danicopan for approximately 40 months. The starting dosage was to be 100 mg TID, and after 2 weeks, the dosage was to be increased to 200 mg TID for participants with body weight ≥ 60 kg or 150 mg TID for participants with body weight < 60 kg. Planned enrollment was approximately 20 participants.

ELIGIBILITY:
Key Inclusion Criteria:

1. At least 12 years of age
2. Completion of the ACH471-201 clinical study OR diagnosed with biopsy-confirmed primary C3G or IC-MPGN
3. If a pre-treatment biopsy is obtained, or if a historical biopsy is available for review, it must have no more than 50% global fibrosis and no more than 50% of glomeruli with cellular crescents
4. Clinical evidence of ongoing disease based on significant proteinuria (defined as ≥500 mg/day of protein in a 24-hour urine) attributable to C3G disease or IC-MPGN in the opinion of the principal investigator (PI), and present prior to study entry and confirmed during Screening
5. If on corticosteroids, anti-hypertensive medications, anti-proteinuric medications (for example, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers), or mycophenolate mofetil, must be on a stable dose for at least 2 weeks prior to screening
6. Female participants must use an acceptable method birth control to prevent pregnancy during the clinical study and for 30 days after the last dose of study medication
7. Male participants must use highly effective birth control with a female partner to prevent pregnancy during the clinical study and for 90 days after the last dose of study medication
8. Must be up-to-date on routine vaccinations, or willing to be brought up-to-date, based on local guidelines
9. Must have access to emergency medical care

Key Exclusion Criteria

1. Have a history of a major organ transplant (for example, heart, lung, kidney, or liver) or hematopoietic stem cell/marrow transplant
2. Have a history or presence of any clinically relevant co-morbidities that would make the participant inappropriate for the study (for example, a comorbidity that is likely to result in deterioration of the participant's condition, affect the participant's safety during the study, or confound the results of the study), in the opinion of the PI
3. Have an eGFR <30 milliliter/minute/1.73 m^2 at the time of screening or at any time over the preceding 4 weeks
4. Is a renal transplant recipient or receiving renal replacement therapy
5. Have other renal diseases that would interfere with the interpretation of the study
6. Have evidence of monoclonal gammopathy of unclear significance, infections, malignancy, autoimmune diseases, or other conditions to which C3G or IC-MPGN is secondary
7. Have been diagnosed with or show evidence of hepatobiliary cholestasis
8. Females who are pregnant, nursing, or planning to become pregnant during the study or within 90 days of ACH-0144471 administration or participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days of ACH-0144471 administration
9. Have a history of febrile illness, a body temperature >38°Celsius, or other evidence of a clinically significant active infection, within 14 days prior to danicopan administration
10. Have evidence of human immunodeficiency virus, hepatitis B infection, or active hepatitis C infection at Screening
11. Have a history of meningococcal infection within the prior year
12. Have a history of hypersensitivity reactions to commonly used antibacterial agents, including beta-lactams, penicillin, aminopenicillins, fluoroquinolones, cephalosporins, and carbapenems, which, in the opinion of the investigator and/or an appropriately qualified immunology or infectious disease expert, would make it difficult to properly provide either empiric antibiotic therapy or treat an active infection.
13. Have participated in a clinical study in which an investigational drug was given within 30 days, or within 5 half-lives of the investigational drug, whichever is longer, prior to the first dose of ACH-0144471
14. Have received eculizumab at any dose or interval within the past 50 days prior to the first dose of ACH-0144471
15. Have received tacrolimus or cyclosporine within 2 weeks of the first dose of ACH-0144471
16. Have a 12-lead electrocardiogram (ECG) with a QT interval Fridericia correction formula >450 millisecond (msec) for males or >470 msec for females, or have ECG findings which, in the opinion of the PI, could put the participant at undue risk
17. Have received any drug known to prolong the corrected QT interval within 2 weeks of the first dose of ACH-0144471 and which, in the opinion of the PI, could put the participant at undue risk
18. Have any of the following laboratory abnormalities at screening:

    * Alanine transaminase > upper limit of normal (ULN)
    * Aspartate aminotransferase > ULN
    * Absolute neutrophil counts <1,000/microliter
    * Total bilirubin >1.5* ULN
    * Indirect bilirubin > ULN
    * Any laboratory abnormality that, in the opinion of the PI, would make the participant inappropriate for the study
19. Unwilling or unable to comply with the study protocol for any reason

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - Clinical Study Site, Birmingham, Alabama
  - Clinical Study Site, Stanford, California
  - Clinical Study Site, New Haven, Connecticut
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Columbus, Ohio
  - Clinical Study Site, Philadelphia, Pennsylvania
- Australia (3):
  - Clinical Study Site, Sydney, New South Wales
  - Clinical Study Site, Brisbane, Queensland
  - Clinical Study Site, Melbourne, Victoria
- Clinical Study Site, Antwerp, Belgium
- Clinical Study Site, Ranica, Italy
- Netherlands (2):
  - Clinical Study Site, Leiden
  - Clinical Study Site, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: SAP, CSR

REFERENCES:
- [Derived] Nester C, Appel GB, Bomback AS, Bouman KP, Cook HT, Daina E, Dixon BP, Rice K, Najafian N, Hui J, Podos SD, Langman CB, Lightstone L, Parikh SV, Pickering MC, Sperati CJ, Trachtman H, Tumlin J, de Vries AP, Wetzels JFM, Remuzzi G. Clinical Outcomes of Patients with C3G or IC-MPGN Treated with the Factor D Inhibitor Danicopan: Final Results from Two Phase 2 Studies. Am J Nephrol. 2022;53(10):687-700. doi: 10.1159/000527167. Epub 2022 Nov 24. PMID 36423588

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: To enroll in the study, participants were required to have a biopsy-confirmed diagnosis of C3 glomerulopathy (C3G) or immune-complex membranoproliferative glomerulonephritis (IC-MPGN).
Period: Overall Study
Arm/Group | Danicopan
Started | 22
Received at Least 1 Dose of Study Drug | 22
Completed | 0
Not Completed | 22
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 1
Not completed — Sponsor's decision to close the study | 18

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug during treatment period.
Arm/Group | Danicopan
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Composite Biopsy Score At End Of Initial 12-Month Treatment Period
Description: The composite biopsy score was based on a score incorporating changes in the activity index, glomerular C3c staining, and glomerular macrophage infiltration at the end of the initial 12 months of treatment. The composite renal biopsy index scoring system ranged from 0 to 21, with higher scores indicating worse outcomes.
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Danicopan
Number analyzed (Participants) | 16
score on a scale
  Baseline | 10.6 (3.59)
  End of 12-Month Initial Treatment Period: number analyzed (Participants) | 9
  End of 12-Month Initial Treatment Period | 8.0 (4.53)
  Change from Baseline: number analyzed (Participants) | 8
  Change from Baseline | -0.9 (1.89)

2. Primary Outcome: Participants With Reduction In Proteinuria At End Of Initial 12-Month Treatment Period
Description: Proteinuria reduction was defined as ≥30% decrease from baseline based on 24-hour urine protein (mg/day).
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Number; unit: participants
Arm/Group | Danicopan
Number analyzed (Participants) | 19
participants | 8

3. Secondary Outcome: Change From Baseline In Proteinuria At End Of Initial 12-Month Treatment Period
Description: Proteinuria was assessed based on 24-hour urine collections at baseline and end of the initial 12-month Treatment Period.
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Danicopan
Number analyzed (Participants) | 22
mg/day
  Baseline | 4252.28 (2684.959)
  End of Initial 12-Month Treatment Period: number analyzed (Participants) | 19
  End of Initial 12-Month Treatment Period | 3512.63 (3335.765)
  Mean Change from Baseline: number analyzed (Participants) | 19
  Mean Change from Baseline | -671.11 (2695.592)

4. Secondary Outcome: Percent Change From Baseline In Proteinuria At End Of Initial 12-Month Treatment Period
Description: Proteinuria was assessed based on 24-hour urine collections at baseline and end of initial 12-month Treatment Period.
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Danicopan
Number analyzed (Participants) | 19
percent change | -17.1 (53.17)

5. Secondary Outcome: Slope Of Estimated Glomerular Filtration Rate (eGFR) From Baseline To End Of Initial 12-Month Treatment Period
Description: Slope of eGFR was estimated using a simple linear regression for each participant, including all data values from baseline until the end of the Initial 12-Month Treatment Period, with eGFR as the dependent variable and time as the independent variable.
Time Frame: End of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2 per month
Arm/Group | Danicopan
Number analyzed (Participants) | 22
mL/min/1.73 m^2 per month | -1.24917 (1.811457)

6. Secondary Outcome: Change From Baseline In eGFR At End Of Initial 12-Month Treatment Period
Description: Change from baseline in eGFR at end of initial 12-Month Treatment Period is presented.
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Danicopan
Number analyzed (Participants) | 22
mL/min/1.73 m^2
  Baseline | 90.692 (35.4939)
  End of Initial 12-Month Treatment Period: number analyzed (Participants) | 20
  End of Initial 12-Month Treatment Period | 81.412 (38.3320)
  Change from Baseline: number analyzed (Participants) | 20
  Change from Baseline | -9.795 (14.3806)

7. Secondary Outcome: Participants With Significant Improvement In eGFR Relative To Baseline At End Of Initial 12-Month Treatment Period
Description: Significant improvement relative to baseline was defined as a ≥ 25% increase from baseline in eGFR.
Time Frame: Baseline, end of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Number; unit: participants
Arm/Group | Danicopan
Number analyzed (Participants) | 20
participants | 0

8. Secondary Outcome: Change From Baseline in eGFR Over 12 Months of Treatment For Participants Meeting eGFR Inclusion Criteria
Description: Participants were eligible for enrollment if inclusion criteria were met including having an eGFR >=30 milliliters (mL)/minute (min)/1.73 square meter (m^2) at the time of screening or at any time over the preceding 4 weeks. This Outcome Measure was registered in case there were participants who were enrolled and ended up not meeting the Eligibility Criteria and was intended to report data for change from baseline in eGFR for only the participants who met the eligibility criteria (that is, participants who did not meet the eligibility criteria would have been excluded from analysis for this Outcome Measure). Since all enrolled participants met the Eligibility Criteria, none of the participants were excluded from this analysis. Therefore, this data is the same data that is presented in Outcome Measure #6 "Change From Baseline In eGFR At End Of Initial 12-Month Treatment Period". Change from baseline in eGFR at end of initial 12-Month Treatment Period is presented.
Time Frame: End of initial 12-Month Treatment Period
Population: All participants who received at least 1 dose of study drug and had analyzable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Danicopan
Number analyzed (Participants) | 22
mL/min/1.73 m^2
  Baseline | 90.692 (35.4939)
  End of Initial 12-Month Treatment Period: number analyzed (Participants) | 20
  End of Initial 12-Month Treatment Period | 81.412 (38.3320)
  Change from Baseline: number analyzed (Participants) | 20
  Change from Baseline | -9.795 (14.3806)

9. Secondary Outcome: Change From Baseline In Measured GFR At The End Of The Initial 12-Month Treatment Period
Description: Data for this Outcome Measure was to be collected where available. None of the sites collected data for this Outcome Measure.
Time Frame: End of initial 12-Month Treatment Period
Population: Analysis was not performed, as data were not collected for this Outcome Measure.
Arm/Group | Danicopan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to 4 weeks after last dose of study drug (up to Week 108)
Arm/Group | Danicopan
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danicopan (N=22)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danicopan (N=22)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Left ventricular failure (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 2 (3)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypertrophy of tongue papillae (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 11 (16)
Oedema peripheral (General disorders) | 8 (15)
Fatigue (General disorders) | 5 (7)
Asthenia (General disorders) | 4 (5)
Influenza like illness (General disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Multiple allergies (Immune system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (11)
Pharyngitis (Infections and infestations) | 6 (6)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (9)
Upper respiratory tract infection (Infections and infestations) | 2 (4)
Urinary tract infection (Infections and infestations) | 2 (4)
Rhinitis (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 1 (2)
Bacteriuria (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Ear lobe infection (Infections and infestations) | 1 (1)
Enterobiasis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 5 (11)
Blood creatinine increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Crystal urine present (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Lipids increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (10)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 6 (13)
Dizziness (Nervous system disorders) | 3 (3)
Migraine (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (2)
Dizziness postural (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hypertensive crisis (Vascular disorders) | 1 (3)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03459443/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03459443/SAP_002.pdf